CLINICAL TRIAL: NCT03089437
Title: The Effects of Prolonged Standing Compared to Prolonged Sitting on Postprandial Lipemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Edward F. Coyle, Dr., University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2016-12-0031
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Metabolic Syndrome; Atherosclerosis
MeSH Terms: conditions — Metabolic Syndrome; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolonged Standing (Experimental): Subject stand for 12 hours. The following day the subject will undergo a high fat tolerance test. Order of sitting/standing will be random and each subject will perform both interventions.
  Interventions: Behavioral: Prolonged Standing
- Prolonged Sitting (Experimental): Subject sit for 12 hours. The following day the subject will undergo a high fat tolerance test. Order of sitting/standing will be random and each subject will perform both interventions.
  Interventions: Behavioral: Prolonged Sitting

INTERVENTIONS:
Behavioral: Prolonged Standing — Subject will stand for 12 hours and undergo a high fat tolerance test the subsequent day
  Arms: Prolonged Standing
Behavioral: Prolonged Sitting — Subject will sit for 12 hours and undergo a high fat tolerance test the subsequent day
  Arms: Prolonged Sitting

SUMMARY:
The effects of 12 hours of prolonged standing will be compared to prolonged standing on a high fat tolerance test the following day. Plasma triglycerides, insulin, and glucose will be measured in a crossover study design.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* heart problems
* coronary artery disease
* hypertension
* respiratory problems
* musculoskeletal problems that prevent prolonged standing or sitting
* obesity
* susceptibility to fainting

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-08-11 (Actual); Study Completion 2018-08-11 (Actual)

PRIMARY OUTCOMES:
Plasma Triglycerides | 6 hours
  The area under the curve for plasma triglycerides from hourly samples during a 6 hour high fat tolerance test
Plasma Insulin | 6 hours
  The area under the curve for plasma insulin from hourly samples during a 6 hour high fat tolerance test
Plasma Glucose | 6 hours
  The area under the curve for plasma glucose from hourly samples during a 6 hour high fat tolerance test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin Human Performance Laboratory, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No